CLINICAL TRIAL: NCT02918734
Title: A Prospective Randomized Controlled Trial Comparing the Endobutton CL BTB Fixation System With Metal Interference Screws in the Femoral Fixation of Patellar Tendon Grafts in Anterior Cruciate Ligament Reconstruction.
Brief Title: Fixation of Patellar Tendon Grafts in Anterior Cruciate Ligament Reconstruction. Endobutton vs Metal Interference Screws
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Rosenborgklinikken (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/993
Record Dates: First submitted 2016-06-20; First posted 2016-09-29 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Knee Injuries
Keywords: Anterior Cruciate Ligament; Bone-Patellar Tendon-Bone Grafting
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endobutton CL BTB (Experimental): Femoral fixation of the BPTB autograft with the Endobutton CL BTB Fixation System.
  Interventions: Device: Endobutton CL BTB
- Metal interference screw (Active Comparator): Femoral fixation of the BPTB autograft with a metal interference screw.
  Interventions: Device: Metal interference screw

INTERVENTIONS:
Device: Endobutton CL BTB — ACL reconstruction with Endobutton CL BTB
  Arms: Endobutton CL BTB
Device: Metal interference screw — ACL reconstruction with metal interference screw
  Arms: Metal interference screw

SUMMARY:
In this randomized controlled trial the investigators will compare the results after primary anterior cruciate ligament (ACL) reconstruction using two different methods for femoral fixation of a bone-patellar tendon-bone (BPTB) autograft. Interference screws have been the standard method for fixing the femoral side of BPTB grafts; however, several pitfalls have been reported. Cortical fixation with the Endobutton CL BTB Fixation System has become available and the clinical results have been described as promising; however, no randomized controlled trials comparing these two femoral fixation methods have been conducted, and there is no published data that confirms that the bone block heals in the tunnel with the newer method.

The aim of our study is to compare the outcome after primary ACL reconstruction with BPTB autografts using the Endobutton CL BTB or metal interference screw for femoral fixation.

DETAILED DESCRIPTION:
Primary anterior cruciate ligament (ACL) reconstructions with bone-patellar tendon-bone (BPTB) autografts have recently been found to have a lower risk of revision compared with hamstring tendon autografts, and BPTB has again become our graft of choice. Interference screws have been the standard method for fixing the femoral side of a BPTB graft; however problems such as damage of the graft and failure due to nonparallel screw placement have been reported. Cortical fixation using a suspensory system has been used for soft-tissue graft fixation for several years, and a corresponding device, the Endobutton CL BTB Fixation System (Smith & Nephew, Inc., Andover, MA, USA), has become available for fixation of bone-tendon-bone grafts. The clinical results after fixation with the Endobutton CL BTB have been described as promising; however, no randomized controlled trials comparing these two fixation methods have been conducted, and there is no published data that confirms that the bone block heals in the tunnel with the newer method.

In this randomized controlled trial, patients undergoing primary ACL reconstruction will be randomized into either an Endobutton group or an interference screw group. The primary aim of the study is to compare these two fixation methods, assessed by patient reported outcomes, laxity, range of motion and muscle strength. Knee related quality of life 2 years after surgery is the primary outcome, measured by the Knee injury and Osteoarthritis Outcome Score (KOOS) subscale "knee related Quality of life (QOL)". Other aims are to see if there is any difference in the integration of the bone block in the femoral tunnel assessed by CT scan, in the risk of developing osteoarthritis assessed by radiographs, or in the risk of a postoperative complication or revision. The patients will be followed up 6 weeks, 6 months, 2 years and 10 years after surgery. CT scan will be performed after 6 months, and radiographs after 2 years and 10 years. In addition details of the rehabilitation will be recorded. Patients undergoing a revision will be followed up but excluded from further comparisons in the study.

Our hypothesis is that there is no difference in the outcome after primary ACL reconstruction with BPTB autografts using the Endobutton CL BTB or metal interference screw for femoral fixation, both with a metal interference screw for the tibial fixation.

ELIGIBILITY:
Inclusion Criteria:

* Primary reconstruction of ACL ruptures
* Surgery at least 6 weeks after injury
* The patient must accept and sign the informed consent form before surgery

Exclusion Criteria:

* Medical indication for using another graft than BPTB autograft (such as history of anterior knee pain or occupations etc. requiring frequent kneeling)
* Previous major surgical procedures in the same knee
* Major additional injuries in the knee (posterior cruciate ligament, lateral collateral ligament, medial collateral ligament, sutured meniscus lesions and major cartilage lesions undergoing cartilage repair)
* Contralateral ACL injury (treated or untreated)
* Present or former serious illness that makes follow-up or rehabilitation difficult (e.g. alcohol or drug abuse, psychiatric disease)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Knee related quality of life | 2 years
  KOOS subscale "knee related Quality of life (QOL)"

SECONDARY OUTCOMES:
Tegner activity scale | 6 months, 2 years, 10 years
Lachman test | 6 weeks, 6 months, 2 years, 10 years
  Anterior translation of the tibia
Muscular strength | 6 months, 2 years, 10 years
  Biodex dynamometer
Bone block integration | 6 months
  CT scan
Osteoarthritis | 2 years, 10 years
  X-ray radiographs
Range of motion | 6 weeks, 6 months, 2 years, 10 years
Knee related quality of life | 6 weeks
  KOOS subscale "knee related Quality of life (QOL)"
Knee related quality of life | 6 months
  KOOS subscale "knee related Quality of life (QOL)"
Knee related quality of life | 10 years
  KOOS subscale "knee related Quality of life (QOL)"
Lysholm functional knee score | 6 weeks, 6 months, 2 years, 10 years
KOOS | 6 weeks, 6 months, 2 years, 10 years
  Knee injury and Osteoarthritis Outcome Score
Pivot shift test | 6 weeks, 6 months, 2 years, 10 years
  Anteroposterior and rotational stability
KT-1000 arthrometer | 6 weeks, 6 months, 2 years, 10 years
  Anterior translation of the tibia

OTHER OUTCOMES:
Complications | Up to 10 years
  Registration
Reoperations | Up to 10 years
  Registration

CONTACTS AND LOCATIONS:
Overall Officials: Jon Olav Drogset, md phd, Principal Investigator — St. Olavs Hospital
Locations (2):
- Norway (2):
  - Department of Orthopedic Surgery, St Olavs Hospital, Trondheim
  - Rosenborgklinikken, Trondheim

IPD SHARING:
Plan to Share IPD: No